CLINICAL TRIAL: NCT00962364
Title: Long-term Evaluation and Follow-up Care of Patients Receiving Intracoronary Bone Marrow-derived Cell Administration for Heart Disease
Brief Title: Long-term Evaluation of Patients Receiving Bone Marrow-derived Cell Administration for Heart Disease
Acronym: BMC registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, A. M. Zeiher, Prof. Dr. Andreas M. Zeiher, Johann Wolfgang Goethe University Hospital
Other Study IDs: 201-01-BMC-Reg
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infarction; Ischemic Cardiomyopathy; Dilated Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma from peripheral blood and bone marrow may me retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AMI: Patients with acute myocardial infarction treated with intracoronary administration of bone marrow derived cells
  Interventions: Biological: autologous bone marrow-derived cells
- ICM: Patients with ischemic cardiomyopathy treated with intracoronary administration of bone marrow derived cells
  Interventions: Biological: autologous bone marrow-derived cells
- DCM: Patients with dilated cardiomyopathy treated with intracoronary administration of bone marrow derived cells
  Interventions: Biological: autologous bone marrow-derived cells

INTERVENTIONS:
Biological: autologous bone marrow-derived cells — autologous bone marrow-derived cells isolated by density gradient centrifugation from 50 ml bone marrow aspirate obtained under local anesthesia

SUMMARY:
This study will provide follow-up information and care of patients who have undergone autologous intracoronary bone marrow cell administration at our institution. Patients are monitored for their response to treatment, progression of heart failure and coronary artery disease, and potential later occurring effects of the administered bone marrow cells.

Patients are eligible for this follow-up study if they have received their first intracoronary bone marrow cell administration for the treatment of cardiac disease at our institution from 2001 ongoing.

Participants are generally seen in the clinic at 12 months and 5 years after cell administration, in the meantime regular yearly telephone contacts are performed until 10 years after cell transplantation.

The detailed description contains the planned procedures that are performed during the clinical visits and, if necessary, at additional contacts.

DETAILED DESCRIPTION:
In detail, the following procedures are performed during the clinical visits and, if necessary, at additional contacts:

* periodic physical examination and blood tests
* non-invasive imaging studies may include echocardiography and magnetic resonance imaging
* electrocardiogram at rest and during treadmill testing (may include spiroergometry testing)
* interrogation of implanted defibrillators / pacemakers for monitoring of arrhythmias

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of heart disease with signs and symptoms of heart failure due to

* acute myocardial infarction or
* ischemic cardiomyopathy with or without previous myocardial infarction or
* dilated cardiomyopathy due to valvular heart disease, hypertensive heart disease, history of myocarditis (no active myocardial infection present)

Exclusion Criteria:

* none, all patients meeting the inclusion criteria will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from heart disease with consecutive signs of heart failure, treated in our clinic or being referred for cell therapy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2001-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of procedural and long-term safety of intracoronary administration of bone marrow cells for the treatment for cardiac disease | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, Prof. Dr, Principal Investigator — Cardiology, Goethe University Frankfurt, Germany
Locations (1):
- Cardiology, Department of Internal Medicine III, Frankfurt, Germany

REFERENCES:
- [Result] Assmus B, Fischer-Rasokat U, Honold J, Seeger FH, Fichtlscherer S, Tonn T, Seifried E, Schachinger V, Dimmeler S, Zeiher AM; TOPCARE-CHD Registry. Transcoronary transplantation of functionally competent BMCs is associated with a decrease in natriuretic peptide serum levels and improved survival of patients with chronic postinfarction heart failure: results of the TOPCARE-CHD Registry. Circ Res. 2007 Apr 27;100(8):1234-41. doi: 10.1161/01.RES.0000264508.47717.6b. Epub 2007 Mar 22. PMID 17379833
- [Derived] Luu B, Leistner DM, Herrmann E, Seeger FH, Honold J, Fichtlscherer S, Zeiher AM, Assmus B. Minute Myocardial Injury as Measured by High-Sensitive Troponin T Serum Levels Predicts the Response to Intracoronary Infusion of Bone Marrow-Derived Mononuclear Cells in Patients With Stable Chronic Post-Infarction Heart Failure: Insights From the TOPCARE-CHD Registry. Circ Res. 2017 Jun 9;120(12):1938-1946. doi: 10.1161/CIRCRESAHA.116.309938. Epub 2017 Mar 28. PMID 28351842
- [Derived] Honold J, Fischer-Rasokat U, Seeger FH, Leistner D, Lotz S, Dimmeler S, Zeiher AM, Assmus B. Impact of intracoronary reinfusion of bone marrow-derived mononuclear progenitor cells on cardiopulmonary exercise capacity in patients with chronic postinfarction heart failure. Clin Res Cardiol. 2013 Sep;102(9):619-25. doi: 10.1007/s00392-013-0574-1. Epub 2013 Apr 24. PMID 23612920
- [Derived] De Rosa S, Seeger FH, Honold J, Fischer-Rasokat U, Lehmann R, Fichtlscherer S, Schachinger V, Dimmeler S, Zeiher AM, Assmus B. Procedural safety and predictors of acute outcome of intracoronary administration of progenitor cells in 775 consecutive procedures performed for acute myocardial infarction or chronic heart failure. Circ Cardiovasc Interv. 2013 Feb;6(1):44-51. doi: 10.1161/CIRCINTERVENTIONS.112.971705. Epub 2013 Jan 29. PMID 23362308
- [Derived] Leistner DM, Seeger FH, Fischer A, Roxe T, Klotsche J, Iekushi K, Seeger T, Assmus B, Honold J, Karakas M, Badenhoop K, Frantz S, Dimmeler S, Zeiher AM. Elevated levels of the mediator of catabolic bone remodeling RANKL in the bone marrow environment link chronic heart failure with osteoporosis. Circ Heart Fail. 2012 Nov;5(6):769-77. doi: 10.1161/CIRCHEARTFAILURE.111.966093. Epub 2012 Aug 30. PMID 22936827
- [Derived] Xu Q, Seeger FH, Castillo J, Iekushi K, Boon RA, Farcas R, Manavski Y, Li YG, Assmus B, Zeiher AM, Dimmeler S. Micro-RNA-34a contributes to the impaired function of bone marrow-derived mononuclear cells from patients with cardiovascular disease. J Am Coll Cardiol. 2012 Jun 5;59(23):2107-17. doi: 10.1016/j.jacc.2012.02.033. PMID 22651868